CLINICAL TRIAL: NCT04775446
Title: Multicentre Observational Study Evaluating the Clinical/Biological Characteristics, Efficacy and Safety of Patients With Malignant Pleural Mesothelioma, Treated by Immunotherapy, in Real Life Setting.
Brief Title: Evaluation of the Clinical/Biological Characteristics, Efficacy and Safety of Patients With Malignant Pleural Mesothelioma, Treated by Immunotherapy
Acronym: MESOIMMUNE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: MESOIMMUNE
Record Dates: First submitted 2021-02-01; First posted 2021-03-01 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Immunotherapy; Pleura; Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with malignant pleural mesothelioma treated with Nivolumab.: Patients with malignant pleural mesothelioma treated with Nivolumab.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data entered in a secure computer database

SUMMARY:
The objective of this multicentre descriptive analysis is to describe the clinical and biological characteristics of patients who have received Programmed cell death 1 (anti-PD1) / (PDL1) Programmed death-ligand 1 (PDL1) immunotherapy outside of a clinical trial in terms of efficacy and safety.

DETAILED DESCRIPTION:
Immunotherapy is now an option in the treatment of malignant pleural mesothelioma. A French study, Mesothelioma Avastin plus Pemetrexed-cisplatin Study 2 (MAPS 2), prospective in 2nd line or more, found 40% and 52% disease control rate with respectively an anti-PD1 antibody or a combo of anti-PD1 and Cytotoxic T-Lymphocyte-Associated protein 4 (anti-CTLA4). Safety was rather good with 14% and 26% grade 3-4 in the Nivolumab and combo group respectively.

Thanks to this trial and data from the literature, Programmed cell death 1 (anti-PD1) / (PDL1) Programmed death-ligand 1 (PDL1) immunotherapy became an option in the treatment of malignant pleural mesothelioma, after validation by a multidisciplinary meeting.

The objective of this multicentre descriptive analysis is to describe the clinical and biological characteristics of patients who have received anti-PD1/PDL1 immunotherapy outside of a clinical trial in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Diagnosis of malignant pleural mesothelioma affirmed by the anatomo-pathological analysis report of a histological sample of the tumour (re-read by MESOPATH).
* Patient who has received at least one injection of anti-PD1 or anti-PDL1 antibodies

Exclusion Criteria:

* Explicit refusal by the patient to collect data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant pleural mesothelioma treated with Nivolumab.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Disease control | 12 weeks
  Disease control rate at 12 weeks

SECONDARY OUTCOMES:
Survival with anti-PD1/PDL1 immunotherapy | 12 weeks
  Overall survival from treatment with anti-PD1/PDL1 immunotherapy
Duration of treatment | 12 weeks
  Duration of treatment with PD1/PDL1 immunotherapy
Survival | 12 weeks
  Overall survival from the start of the first treatment
Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by previous immunotherapy | 12 weeks
  Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by following data: which immunotherapy, date of treatment beginning/end
Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by adverse event | 12 weeks
  Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by following data: numbers of treatment related adverse events from CTCAE v4.0
Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by remarkable event | 12 weeks
  Tolerance of treatment with PD1/PDL1 immunotherapy evaluated by following data: date of best response, date of progression, date of death)
To identify factors predictive of treatment response by immunotherapy in responder patients | 12 weeks
  Identify factors predictive of treatment response by immunotherapy in responder patients by collecting following data: Demographics data, treatment data, and blood test results and histological data
To identify factors predictive of the response of immunotherapy treatment of progressive patients | 12 weeks
  Identify factors predictive of treatment response by immunotherapy of progressive by collecting following data: Demographics data, treatment data, and blood test results and histological data
To identify factors predictive of the response of immunotherapy treatment of all patients | 12 weeks
  Identify factors predictive of treatment response by immunotherapy of all patients by collecting following data: Demographics data, treatment data, and blood test results and histological data
To identify factors predictive of the response of immunotherapy treatment according to follow-up treatment | 12 weeks
  Identify factors predictive of treatment response by immunotherapy according to type of treatment after PD1/PDL1 immunotherapy

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CH Côte basque, Bayonne
  - CHU Brest, Brest
  - CH Cherbourg, Cherbourg
  - CHI Créteil, Créteil
  - CHU Lille, Lille

IPD SHARING:
Plan to Share IPD: No